CLINICAL TRIAL: NCT02974556
Title: Proactive Management of Endoperitoneal Spread in Colonic Cancer
Acronym: PROMENADE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Tommaso Cornali, Prof. Paolo Sammartino, MD Phd, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PROMENADE v1.0
Record Dates: First submitted 2016-11-09; First posted 2016-11-28 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Colon Cancer; Intraperitoneal Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin; Folfox protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard surgical treatment group (Active Comparator): Colon cancer patients (high-risk T3 and T4) without peritoneal or systemic metastases are resected for cure.
  Standard adjuvant systemic chemotherapy (FOLFOX or CAPOX regimens for 6 months) will be reserved in pT3 tumors with poor prognostic factors, pT4 tumor and if lymph-nodes metastases are present. Presence or absence of peritoneal recurrence will be evaluated by MDCT.
  Interventions: Procedure: Standard surgical treatment; Drug: Standard adjuvant systemic chemotherapy
- Proactive management group (Experimental): Colon cancer patients (high-risk T3 and T4) without peritoneal or systemic metastases are resected for cure. Simultaneously patients will undergo infracolic omentectomy, appendectomy, exeresis of the liver round ligament and, in women, a bilateral oophorectomy. At the end of surgical procedure HIPEC will be performed with oxaliplatin 460 mg/m2 and before the beginning of HIPEC an intravenous infusion of 400 mg/m2 of 5-FU and 20 mg/m2 of leucovorin will be administered.
  Standard adjuvant systemic chemotherapy (FOLFOX or CAPOX regimens for 6 months) will be reserved in pT3 tumors with poor prognostic factors, pT4 tumor and if lymph-nodes metastases are present. Presence or absence of peritoneal recurrence will be evaluated by MDCT.
  Interventions: Procedure: Proactive management; Drug: Standard adjuvant systemic chemotherapy

INTERVENTIONS:
Procedure: Standard surgical treatment — Standard surgical treatment (open or laparoscopic techniques) containing at least 12 lymph-nodes for accurate pN staging.
  Arms: Standard surgical treatment group
Procedure: Proactive management — Colon cancer patients (high-risk T3 and T4) without peritoneal or systemic metastases are resected for cure. Simultaneously patients will undergo infracolic omentectomy, appendectomy, exeresis of the liver round ligament and, in women, a bilateral oophorectomy. After positioning three in- and outflow catheters HIPEC perfusion starts with a minimum of 2 L isotonic dialysis fluid at a flow-rate of 1-2 l min and an inflow temperature of 42-43° C with a total of 30 minutes perfusion time. Before the beginning of HIPEC 5-fluouracil and leucovorin will be administrated intravenously to potentiate oxaliplatin activity.
  Arms: Proactive management group
Drug: Standard adjuvant systemic chemotherapy — Adjuvant systemic chemotherapy (according CAPOX or FOLFOX regimens for a total of 6 months) will be reserved in patients with pT3 tumors with poor prognostic factors, in patients with pT4 tumors and when lymph-nodes metastases are present. Presence or absence of peritoneal recurrence will be evaluated by MDCT every six months for the first 24 months and later every year for the next three years in both study arms.
  Other Names: adjuvant capecitabine and oxaliplatin (CAPOX); adjuvant 5-FU and oxaliplatin (FOLFOX)

SUMMARY:
This study aims to determine the oncological effectiveness, compared to standard surgical treatment, of proactive management including target organs for peritoneal spread resection (omentectomy, bilateral adnexectomy, appendectomy, hepatic round ligament resection) and preventive HIPEC (intraperitoneal oxaliplatin with concomitant i.v. 5-fluorouracil/leucovorin) following a curative resection of high-risk ( >/= 5 mm tumor invasion beyond the muscularis propria) T3 and T4 colon cancer in preventing the development of peritoneal metastases. Adjuvant systemic chemotherapy will be reserved in both groups for patients with poor prognostic factors according to Folinic acid/Fluorouracil/Oxaliplatin (FOLFOX) or to Capecitabine/Oxaliplatin (CAPOX) regimens.

Hypothesis:

The hypothesis is that compared to the standard treatment proactive management following curative resection of high-risk T3 and T4 colon cancer will reduce the development of endoperitoneal metastases

DETAILED DESCRIPTION:
Colorectal cancer is one of the leading causes of cancer death in developed countries. Despite recent advances in understanding the molecular pathogenesis and improvements in diagnosis and treatment, more than 1,2 million new cases and 600,000 deaths occur annually worldwide and cure rates remain low for patients with metastatic or recurrent disease. According to reports from the National Cancer Institute, cancer of the colon is a highly treatable and often curable disease when confined to the bowel. Surgery is the primary treatment and results in a cure rate of approximately 50% of the patients; however, recurrence following surgery is a major problem and is often the ultimate cause of death. In colon cancer locoregional recurrence (local recurrence and metachronous peritoneal spread), as the main site of recurrence, is less common (up to 10% of all recurrences) and generally occurs within 3 years of resection. An important concept is the origin of local recurrences and peritoneal metastases that have a common natural history. Specific features of the primary tumor like size and depth of bowel wall invasion (pT3-pT4), which determine a specific clinical evolution (obstruction, perforation with exfoliation of cancer cells) are responsible for endoperitoneal recurrence. Cytoreductive Surgery (CRS) defined as removal of macroscopic abdominal and peritoneal disease combined with Hyperthermic Perioperative Chemotherapy (HIPEC) is the treatment considered standard of care for selected patients with moderate to small volume peritoneal metastases secondary to colorectal cancer. Nevertheless treatment of locoregional recurrence and peritoneal metastases in colon cancer are disappointing first because only 30% of patients can be surgically treated and second because of this 30% only 15- 30% survive 5 years, leaving only 10% of patients with a chance of being cured. Furthermore the economic burden of metastatic colorectal cancer treatment is considerable including the common adverse events associated that increase healthcare resource utilization and considering the addition of biological drugs to standard treatment. An evaluation of CRS combined with HIPEC for peritoneal metastases of colorectal origin in the era of value-based medicine, showed an incremental cost respect to modern chemotherapy regimens of 44,217 US$ for life-year saved, making investment in prevention even more attractive. Despite screening for colorectal cancer in average-risk patients using colonoscopy was associated with a substantially reduced risk of diagnosis with new-onset primary late-stage tumors, colorectal cancer screening remains underused. Analyzing the recent surgical published series, the majority (around 70%), of patients with a diagnosis of colonic cancer operated with curative intent, have a pT3-4 tumor, which is exactly the high-risk class of patients for local recurrence and peritoneal metastases. In this scenario the most effective strategy to combat endoperitoneal recurrence seems prevention. Two previous studies performed in our Institution investigated how a proactive management of peritoneal metastases in colon cancer patients considered at high-risk for peritoneal recurrence according to depth of bowel wall invasion and specific histopathologic features (pT3, pT4 any N, M0, mucinous or signet ring cell pathology) influence outcome. A group of 25 patients for whom inclusion criteria were verified by intraoperative pathologic assessment, were submitted to a "proactive" treatment that included in addition to the standard surgical treatment, a greater omentectomy, appendectomy, exeresis of the liver round ligament and, in post-menopausal women, a bilateral oophorectomy. At the end of the operation, in these patients a HIPEC was performed with oxaliplatin and simultaneous iv infusion of 5-fluorouracil (FU) + leucovorin (LV). Short and long-term results showed that when compared to a control group (50 cases) of similar patients treated only by standard treatment in the same Institution, this group of patients had a statistically significant decreased incidence of peritoneal recurrence (4 vs. 28%) and an increase in overall and disease-free survival rates. These results should obviously validated by larger controlled studies, and this is the aim of the PROMENADE protocol, to verify if the treatment criteria applied in colorectal peritoneal metastases (Surgery combined with HIPEC) could represent a mean of tertiary prevention of endoperitoneal recurrence in high-risk colon cancer. However, simpler application criteria were needed for a large-scale study. For this reason histological typing have not been yet considered an inclusion criteria and will only represent a secondary outcome measure. Furthermore, also considering other experiences, the protocol will use an imaging technique (MDCT) for preoperative selection of high-risk T3 (>/= 5 mm tumor invasion beyond the muscularis propria) and T4 colon cancers, combined in patients with suspected systemic disease after MDCT with functional positron-emission tomography (PET), avoiding the need for an intraoperative frozen-sections pathologic assessment. The results of this study will hopefully confirm the therapeutic rationale that makes microscopic local seeding as the main reason for endoperitoneal recurrence. It will be also important to verify if, as demonstrated in our pilot study, a better loco-regional control of the disease will carry better long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colon cancer or intraperitoneal rectosigmoid cancer with clinical (by CT) high-risk(> 5mm) T3, T4 tumors, any N, M0
* Performance Status (ECOG) 0, 1 or 2
* Signed informed consent

Exclusion Criteria:

* BMI> 30
* Impossibility of an adequate follow-up
* Intra and extraabdominal metastatic disease, multiple colorectal cancer or other malignancies
* Active infections or severe associated medical conditions (ASA IV or V)
* Abnormal bone marrow or renal and liver function indices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of endoperitoneal recurrence at 36 months | 36 months
  The primary endpoint is the incidence of endoperitoneal recurrence at 36 months defined as the proportion of subjects with peritoneal metastases at 36 months from randomization.

SECONDARY OUTCOMES:
disease-free survival (DFS) | 3 years
disease-free survival (DFS) | 5 years
overall survival (OS) | 3 years
overall survival (OS) | 5 years
extraperitoneal (systemic) or liver recurrence rate | 3 years
morbidity rate | 1 month
morbidity rate | 6 months
HIPEC toxicity rate | 1 month
HIPEC toxicity rate | 6 month
EORTC QLQ-C30 Summary Score | 6 months
  The EORTC QLQ-C30 Summary Score range from 0 to 100 and is calculated from the mean of 13 of the 15 QLQ-C30 scales (the Global Quality of Life scale and the Financial Impact scale are not included). Prior to calculating the mean, the symptom scales need to be reversed to obtain a uniform direction of all scales.
  QLQ-C30 Summary Score = (Physical Functioning+ Role Functioning+ Social Functioning+ Emotional Functioning+ Cognitive Functioning+ 100-Fatigue+ 100-Pain+ 100-Nausea_Vomiting+ 100-Dyspnoea+ 100-Sleeping Disturbances+ 100-Appetite Loss+ 100-Constipation+ 100-Diarrhoea)/13
EORTC QLQ-C30 Summary Score | 1 year
  The EORTC QLQ-C30 Summary Score range from 0 to 100 and is calculated from the mean of 13 of the 15 QLQ-C30 scales (the Global Quality of Life scale and the Financial Impact scale are not included). Prior to calculating the mean, the symptom scales need to be reversed to obtain a uniform direction of all scales.
  QLQ-C30 Summary Score = (Physical Functioning+ Role Functioning+ Social Functioning+ Emotional Functioning+ Cognitive Functioning+ 100-Fatigue+ 100-Pain+ 100-Nausea_Vomiting+ 100-Dyspnoea+ 100-Sleeping Disturbances+ 100-Appetite Loss+ 100-Constipation+ 100-Diarrhoea)/13

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Sammartino, MD PhD, Principal Investigator — University of Roma La Sapienza
Locations (8):
- Italy (8):
  - ASST Nord Milano P.O. Città di Sesto S. Giovanni, Milan, PD
  - ASO S. Croce e Carle, Cuneo
  - Azienda Ospedaliera dei Colli, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale di Napoli, Napoli
  - Ospedale di Rimini, Rimini
  - University of Rome Sapienza, Roma
  - Ospedale Sant'Eugenio, Rome
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sammartino P, Biacchi D, Cornali T, Cardi M, Accarpio F, Impagnatiello A, Sollazzo BM, Di Giorgio A. Proactive Management for Gastric, Colorectal and Appendiceal Malignancies: Preventing Peritoneal Metastases with Hyperthermic Intraperitoneal Chemotherapy (HIPEC). Indian J Surg Oncol. 2016 Jun;7(2):215-24. doi: 10.1007/s13193-016-0497-1. Epub 2016 Jan 26. PMID 27065712
- [Background] Sammartino P, Sibio S, Biacchi D, Cardi M, Mingazzini P, Rosati MS, Cornali T, Sollazzo B, Atta JM, Di Giorgio A. Long-term results after proactive management for locoregional control in patients with colonic cancer at high risk of peritoneal metastases. Int J Colorectal Dis. 2014 Sep;29(9):1081-9. doi: 10.1007/s00384-014-1929-4. Epub 2014 Jul 1. PMID 24980687
- [Background] Sammartino P, Sibio S, Accarpio F, Di Giorgio A. Prevention of peritoneal carcinomatosis from colorectal cancer: a critical issue. Ann Surg. 2014 Mar;259(3):e51. doi: 10.1097/SLA.0000000000000372. No abstract available. PMID 24263309
- [Background] Sammartino P, Sibio S, Biacchi D, Cardi M, Accarpio F, Mingazzini P, Rosati MS, Cornali T, Di Giorgio A. Prevention of Peritoneal Metastases from Colon Cancer in High-Risk Patients: Preliminary Results of Surgery plus Prophylactic HIPEC. Gastroenterol Res Pract. 2012;2012:141585. doi: 10.1155/2012/141585. Epub 2012 May 8. PMID 22645605